CLINICAL TRIAL: NCT06798740
Title: Post Market Registry Study of Intracranial Aneurysms Treated With Sugita Clipping Devices
Acronym: T2_PMCF
Status: Recruiting | Type: Observational
Sponsor: Mizuho Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: CE-0005_CIP
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Brain Aneurysm
Keywords: clip; sugita
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aneurysm clip: Patients presenting intracranial aneurysm (ruptured or unruptured) that the physician intends to treat with the Sugita clips.
  Interventions: Device: Sugita Titanium Aneurysm Clip II

INTERVENTIONS:
Device: Sugita Titanium Aneurysm Clip II — Aneurysm clipping is a surgical procedure used to treat brain aneurysms.

SUMMARY:
The objective of this study is to verify the performance and safety of the Sugita Aneurysm Clips devices when used as intended and to identify possible risk factors. Data collected will be used to support the continuing performance and safety of the devices in the post-market use environment in Europe. Subjects who have an intracranial aneurysm that the physician intends to treat with the subject devices will be included in the study. Subjects will be followup as per hospital standard of care for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an intracranial aneurysm (ruptured or unruptured) that can be treated with one of the proposed devices.
* Subject is adult, ≥18 years.
* As per national regulations, subject or subject's legally authorized representative (LAR) has signed written informed consent.
* Subject is willing to comply with scheduled visits and examinations per institutional standard of care.

Exclusion Criteria:

* Subject is currently enrolled in or plans to be enrolled in a concurrent drug or device randomized study.
* Subject has a condition which will not allow him/her to comply with his/her post-procedure follow up per the institutional standard of care (medical condition, subject living abroad and unable to return for follow- up, e.g.).
* Subject does not meet IFU criteria of the subject device.
* Subject is a child, <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have an intracranial aneurysm (ruptured or unruptured) that the physician intends to treat with the subject device(s)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-02-14 (Estimated); Study Completion 2033-02-14 (Estimated)

PRIMARY OUTCOMES:
Rate of permanent aneurysm occlusions | Up to 12 months
  Rate of complete permanent aneurysm occlusions according to Molyneux et al, 2005, where the category of occlusion is selected as "Complete occlusion".

SECONDARY OUTCOMES:
Incidence of adverse events | up to 60 months
  The number and percentage of subjects experiencing any adverse event. Each adverse event type, including severity will be reported.
Change in Modified Rankin Scale | through 60 months
  The mean, standard deviation, median, minimum, maximum, and number of evaluable observations will be reported for baseline and to each follow up visit using descriptive statistics.The absolute change from baseline will be calculated for each subject at follow up visits.
Amount of aneurysm retreatments | through 60 months
  The amount of aneurysm retreatments will be reported as 0, 1 and >=2 retreatments through each follow up visit.
Procedure success rate | within 1 week after clipping
  Rate of successful aneurysm occlusions per Molyneux classification "Complete occlusion" while using a permanent clip. Frequency counts and percentages of subjects, as well as 95% confidence intervals for the percentages will be presented.
Rate of successful applications of temporary clips | Within 1 week after clipping
  Subjects that experience a successful aneurysm occlusion according to Molyneux classification "Complete occlusion" while using temporary clips.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No